CLINICAL TRIAL: NCT06134531
Title: Clinical Study on Evaluating the Safety and Tolerability of Bispecific Antibody MR001 in Patients With Advanced Solid Tumors.
Brief Title: First-In-Human Study of Bispecific Antibody MR001 In Subjects With Advanced Solid Tumors
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Nanfang Hospital, Southern Medical University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NFEC-2023-382
Record Dates: First submitted 2023-10-16; First posted 2023-11-18 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Advanced Solid Tumors

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- MR001 (Experimental): The investigational product is MR001 which will be supplied in glass vials containing 50 mg of Freeze-dried powder. MR001 could be diluted in saline for intravenous (IV) administration.
  Interventions: Drug: MR001

INTERVENTIONS:
Drug: MR001 — Dose Level 1: 0.5 mg/kg Intravenously (IV) Frequency: administered on Day 1 of each cycle (every 3 weeks), 1 cycle
  Dose Level 2: 2 mg/kg Intravenously (IV) Frequency: administered on Day 1 of each cycle (every 3 weeks), 4 cycle
  Dose Level 3: 6 mg/kg Intravenously (IV) Frequency: administered on Day 1 of each cycle (every 3 weeks), 4 cycle
  Dose Level 4: 10 mg/kg Intravenously (IV) Frequency: administered on Day 1 of each cycle (every 3 weeks), 4 cycle
  Dose Level 5: 15 mg/kg Intravenously (IV) Frequency: administered on Day 1 of each cycle (every 3 weeks), 4 cycle
  Dose Level 6: 20 mg/kg Intravenously (IV) Frequency: administered on Day 1 of each cycle (every 3 weeks), 4 cycle
  Other Names: anti-CD4/anti-TGFβ1 bispecific antibody

SUMMARY:
Phase 1 open-label study to evaluate the safety, tolerability and preliminary efficacy of bispecific antibody MR001 and to determine the maximal tolerated dose and designate the recommended phase 2 dose in subjects with locally advanced or metastatic solid cancers.

DETAILED DESCRIPTION:
Phase 1 open-label study to evaluate the safety, tolerability and preliminary efficacy of bispecific antibody MR001 and to determine the maximal tolerated dose and designate the recommended phase 2 dose in subjects with locally advanced or metastatic solid cancers. The study will be conducted in 2 parts: part 1 will involve dose escalation and part 2 will involve expansion of the recommended phase 2 dose.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years old and ≤75 years old (including the critical value);
2. Patients with histologically or cytologically confirmed advanced metastatic solid tumors who have failed standard treatments, are intolerant to standard treatments, or refuse standard treatments;
3. According to RECIST 1.1 criteria, there is at least 1 evaluable target lesion;
4. ECOG score physical status is 0-2;
5. Have appropriate organs and hematopoietic function, and no serious organ dysfunction according to the following laboratory tests:

   Hematology: absolute neutrophil count (ANC) ≥1.5×10e9/L, platelets ≥100×10e9/L, white blood cell count ≥3×10e9/L, hemoglobin ≥90 g/L; Renal function: serum creatinine ≤1.5 times the upper limit of normal (ULN) or creatinine clearance ≥50 mL/min (creatinine clearance using the Cockcroft-Gault formula); Liver function: AST and ALT ≤ 2.5 times ULN, patients with liver metastasis ≤ 5 times ULN; serum bilirubin (TBIL) ≤ 1.5 times ULN; alkaline phosphatase ≤ 1.5 times ULN, patients with liver metastasis or bone metastasis ≤ 5 times ULN ; Coagulation function: international normalized rate (INR) or activated partial thromboplastin time (APTT) ≤ 1.5 times ULN;
6. CD4+T lymphocyte count >350 cells/μL;
7. Expected survival ≥3 months;
8. No birth plans within 2 weeks before screening and 3 months after the end of the trial and agree to take effective non-drug contraceptive measures during the trial;
9. Voluntarily participate in the trial and sign the informed consent form.

Exclusion Criteria:

1. Those who are allergic to trial drugs or excipients;
2. Subjects with uncontrolled active brain metastasis or meningeal metastasis: those who need to use any radiation, surgery or drug treatment (including steroids, anticonvulsant drugs, etc.) to control metastasis symptoms 1 month before screening are not allowed Enrollment, patients with stable brain metastases can be enrolled;
3. Those who have suffered from autoimmune diseases in the past and need to use glucocorticoids or immunosuppressive drugs;
4. Uncontrolled comorbidities or cancer pain;
5. Hypertension that remains uncontrollable after drug treatment (systolic blood pressure >170 mmHg or diastolic blood pressure >100 mmHg);
6. Those with a history of severe heart disease, such as: a history of acute myocardial infarction or coronary angioplasty or stent implantation within 12 months, unstable angina, myocarditis, chronic heart failure ≥ grade III (New York, USA) Heart Association standards), or those with a history of QT interval prolongation (>470 ms for women; >450 ms for men) or a history of severe arrhythmia as shown by electrocardiogram;
7. Those with a history of severe kidney disease, such as chronic nephritis, renal insufficiency, etc.;
8. There is currently an uncontrolled active infection;
9. Active hepatitis B (HBsAg positive, and peripheral blood HBV DNA titer test ≥1×10e3 IU/mL), hepatitis C, syphilis-specific antibodies and human immunodeficiency virus (HIV) antibody screening Patients with positive test results;
10. Other malignant tumors occurred within 5 years before screening, except for cervical cancer in situ, cutaneous squamous cell carcinoma or basal cell carcinoma that has been previously treated for radical treatment;
11. Those who have received the COVID-19 vaccine within 28 days before screening or have received other vaccines within 3 months before screening or plan to receive vaccines during the trial;
12. Subjects who received systemic steroid treatment within 14 days before the first dose and were judged by the investigator to need long-term systemic steroid treatment during treatment (except for inhaled or topical use, physiological replacement dose);
13. Participated in any other interventional clinical trial within 28 days before the first dose;
14. Received blood transfusion and/or colony-stimulating factor-related treatment within 28 days before the first dose;
15. Those who have received major surgical and/or anti-tumor treatments (including but not limited to chemotherapy, radiotherapy, targeted and immunotherapy, etc.) within 28 days before the first dose, and have failed to recover from the toxicity of these interventions (according to NCI-CTCAE version 5.0 toxicity has not returned to ≤ grade 1), except for alopecia;
16. Women preparing for pregnancy, pregnancy, and lactation;
17. Any other circumstances that the researcher believes may increase the risk to the subjects or interfere with the results of the trial, and who are deemed unsuitable to enter this trial.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Estimated)
Dates: Start 2023-11 (Estimated); Primary Completion 2026-07 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Incidence of treatment-emergent adverse events, and serious adverse events | 12 months
  Safety profile of MR001
Dose Limited Toxicity (DLT) and Maximum Tolerated Dose (MTD) | 12 months
  Determine the DLT and MTD and designate a recommended phase 2 dose (RP2D)

SECONDARY OUTCOMES:
Peak Time (Tmax) of MR001 | 12 months
  Determine the Tmax of MR001
Maximum Plasma Concentration (Cmax) of MR001 | 12 months
  Determine the Cmax of MR001
Area under the Concentration versus Time Curve (AUC) of MR001 | 12 months
  Determine the AUC(0-t) and AUC(0-∞) of MR001
Elimination of Half-life (t1/2) of MR001 | 12 months
  Determine the t1/2 of MR001
Clearance (CL) of MR001 | 12 months
  Determine the CL of MR001
Volume of Distribution (Vd) of MR001 | 12 months
  Determine the Vd of MR001
Objective Response Rate (ORR) | 12 months
  ORR in accordance with Response Evaluation Criteria in Solid Tumors (RECIST) Version 1.1 and modified RECIST guidelines for immunotherapy trials (iRECIST).
Progression Free Survival (PFS) | 12 months
  Progression-free Survival (PFS) by RECIST Version 1.1 and iRECIST.
Overall Survival (OS) | 12 months
  Overall Survival (OS) by RECIST Version 1.1 and iRECIST.
Duration of Response (DOR) | 12 months
  Duration of Response (DOR) by RECIST Version 1.1 and iRECIST.
Disease Control Rate (DCR) | 12 months
  Disease Control Rate (DCR) by RECIST Version 1.1 and iRECIST.
Anti-drug Antibody (ADA) | 12 months
  Determine the Anti-MR001 antibody in the plasma

CONTACTS AND LOCATIONS:
Overall Officials: Guoxin Li, MD, Principal Investigator — Nanfang Hospital, Southern Medical University
Locations (1):
- Nanfang Hospital, Southern Medical University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Li S, Liu M, Do MH, Chou C, Stamatiades EG, Nixon BG, Shi W, Zhang X, Li P, Gao S, Capistrano KJ, Xu H, Cheung NV, Li MO. Cancer immunotherapy via targeted TGF-beta signalling blockade in TH cells. Nature. 2020 Nov;587(7832):121-125. doi: 10.1038/s41586-020-2850-3. Epub 2020 Oct 21. PMID 33087933
- [Result] Liu M, Kuo F, Capistrano KJ, Kang D, Nixon BG, Shi W, Chou C, Do MH, Stamatiades EG, Gao S, Li S, Chen Y, Hsieh JJ, Hakimi AA, Taniuchi I, Chan TA, Li MO. TGF-beta suppresses type 2 immunity to cancer. Nature. 2020 Nov;587(7832):115-120. doi: 10.1038/s41586-020-2836-1. Epub 2020 Oct 21. PMID 33087928